CLINICAL TRIAL: NCT04380298
Title: Effects of Pre-emptive Scalp Infiltration With Low-dose Ketorolac and Ropivacaine for Postoperative Pain Relief After Elective Supratentorial Craniotomy (PAINLESS): a Randomized Controlled Pilot Trial
Brief Title: Effects of Pre-emptive Scalp Infiltration With Low-dose Ketorolac and Ropivacaine for Postoperative Pain
Acronym: PAINLESS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY-2018-034-02-7
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Pain; Supratentorial Brain Tumor
Keywords: Pre-emptive Scalp Infiltration; Ketorolac; Postoperative Pain; Supratentorial Craniotomy; A pilot Study
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ketorolac; Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ketorolac group (Experimental): Patients assigned to the ketorolac group will receive pre-emptive scalp infiltration with 30ml of local infiltration solution containing 60 mg ropivacaine, 6 mg ketorolac and 0.1mg epinephrine.
  Interventions: Drug: Ketorolac; Drug: Ropivacaine; Drug: Epinephrine
- The control group (Active Comparator): In the control group, preoperative peri-incisional scalpinfiltration will be performed using 30ml of 60 mgropivacaine and 0.1mg epinephrine.
  Interventions: Drug: Ropivacaine; Drug: Epinephrine

INTERVENTIONS:
Drug: Ketorolac — 30ml of local infiltration solution containing 60mg ropivacaine
  Arms: The ketorolac group
Drug: Ropivacaine — 30ml of local infiltration solution containing 6mg ketorolac
Drug: Epinephrine — 30ml of local infiltration solution containing 0.1mg epinephrine

SUMMARY:
The PAINLESS study is a single-center, prospective, randomized, open-label, blinded-endpoint (PROBE) controlled clinical pilot study to compare the efficacy and safety of pre-emptive scalp infiltration with ropivacaine plus ketorolac and ropivacaine alone for postoperative pain relief in adults undergoing elective supratentorial craniotomies.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective supratentorial tumour resection;
* Planned general anaesthesia;
* American Society of Anesthesiologists (ASA) physical status I - II;
* Age ranging from 18 to 65 years old;
* Participates required to fix their head in a head clamp intraoperatively;
* Participates with an anticipated awake within 2 hours after surgery.

Exclusion Criteria:

* Allergy/intolerance to study drugs including anesthetic drugs, ketorolac and epinephrine;
* Expected delayed extubation or no plan to extubate;
* History of neurosurgeries;
* Long-term use of analgesics and sedatives (more than 2 weeks)
* Receiving any painkiller within 24 h before the operation;
* Extreme body mass index (BMI) (less than 15 or more than 35);
* Patients with impaired cardiopulmonary;
* Patients with impaired renal function;
* Patients with impaired hepatic function;
* History of chronic headache;
* Patients with cognitive deficit;
* Patients with intellectual disability;
* Patients with uncontrolled epilepsy;
* Patients with psychiatric disorders;
* Difficulties in using PCA device
* Difficulties in understanding the use of numeral rating scale (NRS) ;
* Patients with suspected intracranial hypertension;
* Pregnant or at breastfeeding;
* Infection at the incisional site;
* History of radiation therapy and chemotherapy preoperatively
* With great likelihood of postoperative radiation therapy and chemotherapy based on preoperative imaging.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
cumulative doses of patient-controlled analgesia (PCA) sufentanil consumption | 0 to 48 hours postoperatively
  cumulative doses of patient-controlled analgesia (PCA) butorphanol consumption from 0 to 48 h postoperatively The primary outcome measure will be cumulative doses of PCA butorphanol consumption from 0 to 48 h postoperatively

SECONDARY OUTCOMES:
The time to first request for PCA sufentanil | 0 to 48 hours postoperatively
  The time to first request for patient-controlled analgesia
frequency of pressing PCA pump | Within 48hours postoperatively
  frequency of pressing PCA pump
numeral rating scale (NRS) Score | at 2 hours, 4 hours, 8 hours, 24 hours, 48 hours postoperatively
  0 for"no pain" and 10 for "pain as severe as you can imagine"
Pain control satisfaction score (PCSS) postoperatively | at 24 hours and 48 hours post-operation
  0 for unsatisfactory and 10 for very satisfactory
Ramsay sedation score (RSS) | at 2 hours, 4 hours, 8 hours, 24 hours and 48 hours postoperatively
  1: Anxious, agitated, restless; Ramsey 2: Cooperative, oriented, tranquil; Ramsey 3: Responsive to commands only If Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to lightglabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to lightglabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.
pulse oxygen saturation(SpO2) | 1 minutes before anesthesia induction, 1 minutes after anesthesia induction, 1 minutes after scalp infiltration, at the beginning of skull drilling, mater cutting and skin closure and at 2hours, 4 hours, 8 hours , 24 hours and 48 hours postoperatively
mean arterial blood pressure(MAP) | 1 minutes before anesthesia induction, 1 minutes after anesthesia induction, 1 minutes after scalp infiltration, at the beginning of skull drilling, mater cutting and skin closure and at 2hours, 4 hours, 8 hours , 24 hours and 48 hours postoperatively
heart rate(HR) | 1 minutes before anesthesia induction, 1 minutes after anesthesia induction, 1 minutes after scalp infiltration, at the beginning of skull drilling, mater cutting and skin closure and at 2hours, 4 hours, 8 hours , 24 hours and 48 hours postoperatively
respiratory rate(RR) | 1 minutes before anesthesia induction, 1 minutes after anesthesia induction, 1 minutes after scalp infiltration, at the beginning of skull drilling, mater cutting and skin closure and at 2hours, 4 hours, 8 hours , 24 hours and 48 hours postope
Length of hospital stay | Length of hospital stay, an arverage of 2 weeks
postoperative nausea and vomiting(PONV) | within 48 hours postoperatively
The presence of respiratory depression | within 48 hours postoperatively
  respiratory rate <10 breaths per minute or SpO2 was<90 %
The incidence of haematoma, wound infection or gastric ulcers | during hospitalization, within 2 weeks postoperatively
  side effects

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Song J, Li L, Yu P, Gao T, Liu K. Preemptive scalp infiltration with 0.5% ropivacaine and 1% lidocaine reduces postoperative pain after craniotomy. Acta Neurochir (Wien). 2015 Jun;157(6):993-8. doi: 10.1007/s00701-015-2394-8. Epub 2015 Apr 7. PMID 25845547
- [Background] Kerr DR, Kohan L. Local infiltration analgesia: a technique for the control of acute postoperative pain following knee and hip surgery: a case study of 325 patients. Acta Orthop. 2008 Apr;79(2):174-83. doi: 10.1080/17453670710014950. PMID 18484242
- [Background] Niemelainen M, Kalliovalkama J, Aho AJ, Moilanen T, Eskelinen A. Single periarticular local infiltration analgesia reduces opiate consumption until 48 hours after total knee arthroplasty. A randomized placebo-controlled trial involving 56 patients. Acta Orthop. 2014 Dec;85(6):614-9. doi: 10.3109/17453674.2014.961399. Epub 2014 Sep 19. PMID 25238439
- [Background] Andersen KV, Nikolajsen L, Haraldsted V, Odgaard A, Soballe K. Local infiltration analgesia for total knee arthroplasty: should ketorolac be added? Br J Anaesth. 2013 Aug;111(2):242-8. doi: 10.1093/bja/aet030. Epub 2013 Mar 20. PMID 23514638